CLINICAL TRIAL: NCT05212844
Title: Utilizing the McKenzie Method of Mechanical Diagnosis and Therapy for Management of Cervicogenic Headache: A Prospective Case Series
Brief Title: McKenzie Method of Mechanical Diagnosis and Therapy for Management of Cervicogenic Headache: A Prospective Case Series
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Faith Regional Health Services (Other)
Collaborators: Tufts University (Other); D'Youville College (Other)
Responsible Party: Principal Investigator, Lan Lin Pu, Principal Investigator, Faith Regional Health Services
Other Study IDs: 081468
Record Dates: First submitted 2021-12-17; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic Headache; McKenzie; Neck Pain
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Musculoskeletal Physical Therapy — Therapeutic exercise and manual physical therapy based on the individual response to end range repeated movements.
  Other Names: Mechanical Diagnosis and Treatment

SUMMARY:
The goal of this study is to examine the effectiveness the Mechanical Diagnosis and Therapy (MDT) approach for the management patients with neck related headache that are referred to a hospital based out-patient physical therapy clinic.

Background: Headache conditions are among the most common complaints causing people to seek medical care. An estimated 14 billion dollars are spent annually on treating headaches. Neck related headache is characterized by pain which comes from the cervical spine (neck) and could be referred to the head and/or face. CGH is frequently managed clinically utilizing an MDT approach however to date there is limited research available examining the effectiveness of this intervention type in a population with CGH.

DETAILED DESCRIPTION:
Objective: The goal of this case-series is to examine the effectiveness the Mechanical Diagnosis and Therapy (MDT) approach for the management patients with cervicogenic headache referred to a hospital based out-patient physical therapy clinic.

Design: Prospective consecutive case series.

Background: Headache conditions are among the most common complaints causing people to seek medical care. An estimated 14 billion dollars are spent annually on treating headaches. Cervicogenic headache (CGH) is described as a secondary type of headache characterized by pain which emanates from the cervical spine and is potentially referred to one or more regions of the head and/or face. CGH is frequently managed clinically utilizing an MDT approach however to date there is limited research available examining the effectiveness of this intervention type in a population with CGH.

Study Selection Criteria: Convenience sampling will be utilized. Subjects diagnosed with CGH and meeting inclusion criteria will be recruited from a population of patients referred by their physician to a hospital based out-patient physical therapy clinic for treatment.

Procedures: Subjects meeting inclusion criteria will be evaluated, classified, and receive interventions based on the MDT approach. Outcome measures utilized will include the Neck Disability Index (NDI), Numeric Pain Rating Scale (NRS), and Headache Disability Index (HDI) will be completed at baseline, visit 5, and visit 10 or discharge, whichever comes first.

Data Management: Descriptive statistics will be used to describe sample characteristics. A repeated measures ANOVA will be utilized to identify changes in group means.

Key Words: Cervicogenic Headache, Mechanical Diagnosis and Treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-70
* During the physical therapy examination, it is found that movements, static positions, or postures affect the patient headache symptoms.
* Pain presents as unilateral or bilateral head/neck pain and/or stiffness
* Headache frequency at least 1x/week
* Headache symptoms are present for at least 3 months
* Dizziness and/or tinnitus affected by neck movements or positions
* Patient has been previously screened for their headache symptoms by their MD

Exclusion Criteria:

* Headache is determined to be of non-cervical origin including migraine, cluster headache, tension-type headache
* Malignancy/infection
* Cranial or cervical vascular disorder
* Substance use or withdrawal
* Acute Post cervical surgery
* Psychosis/psychiatric disorder/post-traumatic stress disorder
* Received nerve block or Botox injections during therapy
* Vertigo with nystagmus is present
* Involved in litigation related to headache complaints

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of 15-20 subjects is expected. Subjects referred to physical therapy by their physician and meeting the inclusion criteria will be recruited for participation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Neck Disability Index (NDI) Scores to Discharge | Baseline and 6 weeks
  The NDI measures the patient perceived level of function related to neck pain. The NDI is a 10 item questionnaire scored from 0-50 with higher scores indicating greater levels of disability.
Change from Baseline in Numeric Pain Rating Scale (NPRS) Scores to discharge | Baseline and 6 weeks
  The NPRS is an 11 item numeric scale that provides a patient rating of neck pain and headache symptoms. The scales corelates with a score of 0 indicating "no pain" and 10 indicating the "worst pain imaginable".
Change from Baseline in Headache Disability Index (HDI) Scores to Discharge | Baseline and 6 weeks
  The HDI measures the patient perceived level of pain and disability related to headache symptoms. The HDI is a 25 item questionnaire scored from 0-100 with a higher score indicating a greater level of disability related to the patient headache symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ronal Schenk, PhD, Study Director — Tufts University
Locations (1):
- Faith Regional Rehabilitation Therapies, Norfolk, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided
If data is shared it would be deidentified data reported in aggregate format only.

REFERENCES:
- [Background] Hu XH, Markson LE, Lipton RB, Stewart WF, Berger ML. Burden of migraine in the United States: disability and economic costs. Arch Intern Med. 1999 Apr 26;159(8):813-8. doi: 10.1001/archinte.159.8.813. PMID 10219926
- [Background] Headache Classification Subcommittee of the International Headache Society. The International Classification of Headache Disorders: 2nd edition. Cephalalgia. 2004;24 Suppl 1:9-160. doi: 10.1111/j.1468-2982.2003.00824.x. No abstract available. PMID 14979299
- [Background] Jull G, Barrett C, Magee R, Ho P. Further clinical clarification of the muscle dysfunction in cervical headache. Cephalalgia. 1999 Apr;19(3):179-85. doi: 10.1046/j.1468-2982.1999.1903179.x. PMID 10234466
- [Background] Jull G, Kristjansson E, Dall'Alba P. Impairment in the cervical flexors: a comparison of whiplash and insidious onset neck pain patients. Man Ther. 2004 May;9(2):89-94. doi: 10.1016/S1356-689X(03)00086-9. PMID 15040968
- [Background] Nilsson N. A randomized controlled trial of the effect of spinal manipulation in the treatment of cervicogenic headache. J Manipulative Physiol Ther. 1995 Sep;18(7):435-40. PMID 8568424
- [Background] Page P. Cervicogenic headaches: an evidence-led approach to clinical management. Int J Sports Phys Ther. 2011 Sep;6(3):254-66. PMID 22034615